CLINICAL TRIAL: NCT05956834
Title: A Multi-Modal Remote Monitoring Platform for Frontotemporal Lobar Degeneration (FTLD) Syndromes
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other); BioSensics (Industry)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Other Study IDs: IRB00341607
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PSP; CBD; Progressive Supranuclear Palsy; FTD; Corticobasal Degeneration; Frontotemporal Dementia; Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Frontotemporal Dementia; Frontotemporal Lobar Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PAMSys — Wearable accelerometer and gyroscope for measuring movement
Device: LEGSys — Wearable accelerometer and gyroscope for measuring movement

SUMMARY:
The primary objective of this study is to enroll an observational cohort of approximately 60 patients with PSP over the course of 24 months using a multicenter study design and to follow each of them for 12 months.

The secondary objective of this study is to develop a robust solution for multi-modal remote monitoring of motor symptoms and function in PSP that can be applied to other Frontotemporal lobar degeneration (FTLD) syndromes.

DETAILED DESCRIPTION:
The goal of this project is to develop a robust multi-modal platform for remote monitoring of motor symptoms and cognitive function in FTLD syndromes using wearable sensors and mobile health technology to assess speech, motor, and cognitive functions. The solution will be validated in Progressive Supranuclear Palsy (PSP) by collecting longitudinal data from 60 PSP individuals with PSP. Enrollment will take place over a period of 24 months, though each participant will only be followed for 12 months for data collection. The participants will consist of adult volunteers from two leading CurePSP Centers of Care located at the Atypical Parkinsonism Center at Johns Hopkins Hospital in Baltimore, MD and Massachusetts General Hospital (MGH) in Boston, MA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of possible or probable PSP as defined by the 2017 MDS criteria
* Fluent in reading and speaking English and capable of providing informed consent based on the principal investigator's judgement
* Able to walk 10 feet unassisted at the time of initial enrollment
* Must have a caregiver or study partner who is willing and able to assist with all study-related procedures

Exclusion Criteria:

* Any neurological, medical, or psychiatric condition that would preclude participation in study activities based on the investigator's judgment.
* A history of frequent falls defined as more than 5 falls per month, or who require a walker to ambulate safely at baseline will not be eligible to participate in the study.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study intends to enroll a diverse population of individuals representative of the general PSP population. There are no restrictions based upon race or ethnic origin. This study will recruit both male and female participants aged 40 years or older with a clinical diagnosis of possible or probable PSP phenotype as defined by the 2017 MDS criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 12 months
  Feasibility will be defined by the number of participants who complete the 12 month study and who wear their PAMSys pendant sensors at least 16 hours/day for at least 75% of the designated sensor days (7 days per month).

SECONDARY OUTCOMES:
PSPRS | 12 months
  The Progressive Supranuclear Palsy Rating Scale will be administered in-person every 3 months. The PSPRS is a 28 item scale with a total score of 0-100 where lower scores are less affected.
Cortical Basal ganglia Functional Scale (CBFS) | 12 months
  The Cortical Basal ganglia Functional Scale (CBFS) will be performed every 3 months. The CBFS is a 31 item scale, with a total of 124 possible points, where a lower score is less affected.
PSP Quality of Life scale (PSP QoL) | 12 months
  The PSP Quality of Life scale will be performed every 3 months. The PSP-QoL is a 45 item scale, with a possible scale of 0-100 with lower scores less affected.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after completion of the study and for 24 months.